CLINICAL TRIAL: NCT05771714
Title: Clinical Performance Evaluation of the CareSuperb™ COVID-19 Antigen Home Test
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Cancel study
Sponsor: AccessBio, Inc. (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CT-22255-PR
Record Dates: First submitted 2023-03-14; First posted 2023-03-16 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: COVID-19
Keywords: SARS-CoV-2, COVID-19, Home Test
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: This is an open label, prospective, randomized clinical agreement study to evaluate the sensitivity and specificity of the CareSuperb™ COVID-19 Antigen Home Test when a lay person conducts the test on themselves, or another study participant, as compared to EUA authorized high sensitivity RT-PCR comparator tests.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- individuals ages 14 years and older (Experimental): This kit is intended for non-prescription home use with self-collected direct anterior nares swab samples from individuals ages 14 years and older.
  Interventions: Device: CareSuperb COVID-19 Antigen Home Test Kit
- individuals aged 2 to 13 years (Experimental): This kit is intended for non-prescription home use with self-collected direct anterior nares swab samples.
  If the subject is under the age of 14, an adult lay-user will collect the sample.
  Interventions: Device: CareSuperb COVID-19 Antigen Home Test Kit

INTERVENTIONS:
Device: CareSuperb COVID-19 Antigen Home Test Kit — At home COVID-19 antigen test kit

SUMMARY:
The purpose of this study is to evaluate the accuracy of the CareSuperb™ COVID-19 Antigen Home Test (sensitivity and specificity) in a simulated home use environment when compared to the Roche cobas SARS-CoV-2 (EUA200009), Hologic Panther Fusion SARS-CoV-2 (EUA200014), and Roche cobas SARS-CoV-2 Nucleic acid test for use on the cobas Liat System (EUA210388) high sensitivity Emergency Use Authorization (EUA) SARS-CoV-2 RT-PCR assays.

DETAILED DESCRIPTION:
This is an open label, prospective, randomized clinical agreement study to evaluate the sensitivity and specificity of the CareSuperb™ COVID-19 Antigen Home Test when a lay person conducts the test on themselves, or another study participant, as compared to EUA authorized high sensitivity RT-PCR comparator tests.

Patients presenting to the study site for COVID-19 testing who have signed the informed consent and assent, if applicable, and who meet the eligibility criteria will be enrolled in the study. Upon enrollment, the subject will be assigned a unique subject identification (ID) number. After obtaining relevant demographic and medical information, testing will ensue.

The first sample, collected by the clinical research staff, will be for the standard of care (SOC). Results of the SOC test will be used for subject treatment and management. To mitigate any potential bias which may affect the subject's visual interpretation of the CareSuperb™ test result, the study staff will not provide the SOC test results to the subject until after the results of the CareSuperb™ test are read by the subject.

There will be a 15-minute minimum wait period prior to the collection of the second anterior nares swab sample and an additional 15-minute minimum wait period between the second and third sample collection.

For Even numbered subjects, the second sample, collected by a study staff member, will be used for the RT-PCR comparator tests. The third sample will be collected and tested by the lay user, using the CareSuperb™ COVID-19 Antigen Home Test.

For Odd numbered subjects, the second sample will be collected and tested by the lay user using the CareSuperb™ COVID-19 Antigen Home Test. The third sample will be collected by a study staff member and will be used for the RT-PCR comparator tests.

The clinical study staff member will photograph each subject's test cartridge, labeled with their corresponding subject ID number. Additionally, the study staff member will record whether or not they agree with the test result's interpretation by the subject, and if not, why.

The RT-PCR sample will be placed in the provided viral transport medium (VTM) vial and stored in a -70°C freezer until ready for shipment to the central lab.

The comparator samples for RT-PCR testing will be shipped to the central lab weekly, unless directed otherwise by either the sponsor or the Clinical Research Organization (CRO). Specimens should be shipped on dry ice for next day delivery, avoiding weekend delivery. RT-PCR testing will be performed by the central lab and residual samples will be stored. The central lab will report both the qualitative results for each sample, i.e., positive or negative for COVID-19, and the cycle threshold (Ct) value for all positive samples.

ELIGIBILITY:
Inclusion Criteria:

1. An Institutional Review Board (IRB) approved informed consent and assent (if applicable) is signed and dated prior to any study related activities.
2. Male and female subjects 2 years of age and older, presenting to the site seeking COVID-19 testing. If symptomatic, symptom onset must be within 5 days of enrollment into the study.
3. Subject is willing to provide a self-collected nasal swab sample. (If under the age of 14, the sample will be collected by an adult lay user.)
4. Subject is willing to have nasal swabs collected by a member of the study staff.
5. Subject agrees to complete all aspects of the study.

Exclusion Criteria:

1. Subject is undergoing treatment currently and/or within the past 30 days of study enrollment with medication to treat SARS-CoV-2, which may include but is not limited to Paxlovid, Remdesivir.
2. Subject is receiving convalescent plasma therapy for SARS-CoV-2.
3. Subject used a nasal wash or nasal aspirate treatment on enrollment day.
4. Subject is currently receiving or has received within the past thirty (30) days of the study visit an experimental biologic treatment or therapy, or drug.
5. Subjects who report or whose clinical status or history indicates that they take biotin >10 mg per day.
6. Subjects who previously enrolled in this study.
7. Subject has a visual impairment that cannot be restored with glasses or contact lenses.
8. Subject has prior medical or laboratory training.
9. Subject has prior knowledge of their current COVID-19 infection status.
10. Subject with a history of frequent or difficult to control nosebleeds within the last fourteen (14) days.
11. Subject has received a positive COVID-19 test result within the past sixty (60) days.

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 786 (Actual)
Dates: Start 2023-01-09 (Actual); Primary Completion 2023-05-11 (Actual); Study Completion 2023-05-11 (Actual)

PRIMARY OUTCOMES:
Positive percent agreement with sensitivity | within two weeks of study enrollment
  Compare the positive result between CareSuperb COVID-19 Ag Home Test and three RT-PCR comparators.
Negative percent agreement with specificity | within two weeks of study enrollment
  Compare the negative result between CareSuperb COVID-19 Ag Home Test and three RT-PCR comparators.

CONTACTS AND LOCATIONS:
Overall Officials: Hyeonsuk Kim, Study Director — Access Bio
Locations (1):
- L&A Morales Healthcare, Inc., Miami, Florida, United States